CLINICAL TRIAL: NCT05114213
Title: MR-Guided Adaptive Stereotactic Body Radiotherapy (SBRT) of Primary Tumor for Pain Control in Metastatic Pancreatic Ductal Adenocarcinoma (mPDAC) - a Randomized, Controlled Clinical Study
Brief Title: MR-Guided Adaptive SBRT of Primary Tumor for Pain Control in Metastatic PDAC
Acronym: MASPAC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual, close out in November 2025
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Heidelberg University (Other); University of Zurich (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Dipl.-Phys. Maximilian Niyazi, Vice Chair, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-973
Record Dates: First submitted 2021-10-16; First posted 2021-11-09 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Pancreatic Cancer
Keywords: metastatic pancreatic cancer; SBRT; MR linac; chemotherapy; pain control
MeSH Terms: conditions — Pancreatic Neoplasms; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: SBRT (Experimental): mPDAC patients not progressing after 8 weeks of standard of care systemic therapy (SoC-CT: minimum doublet chemotherapy). The primary tumor is treated with SBRT (6.6Gy x 5) on a MR-LINAC in breath-hold technique. For this purpose, daily adaptive planning is performed aiming to maintain stringent dose constraints for organs at risk (duodenum / stomach / bowel / kidney). Chemotherapy will be continued after SBRT.
  Interventions: Radiation: SBRT; Drug: SOC chemotherapy
- Arm B: SOC (Active Comparator): Continuing SoC-CT (according to clinical routine appr. 2 weeks after the previous cycle) without SBRT.
  Interventions: Drug: SOC chemotherapy

INTERVENTIONS:
Radiation: SBRT — online adaptive MR-guided hypofractionated stereotactic radiotherapy
  Other Names: oMRgRT
  Arms: Arm A: SBRT
Drug: SOC chemotherapy — The chemotherapy is given according to current standard of care, consisting of in minimum doublet - chemotherapy and excluding monotherapy regimens.

SUMMARY:
The MASPAC trial investigates the added benefit of MR-guided adaptive SBRT of the primary tumor embedded between standard chemotherapy cycles for pain control and prevention of pain in patients with metastatic PDAC (mPDAC).

DETAILED DESCRIPTION:
Patients not progressing after 8 weeks of standard of care systemic therapy (SoC-CT: minimum doublet chemotherapy) will be included and randomized between arm A, receiving MR-guided adaptive SBRT of the primary tumor combined with continuation of SoC-CT, and arm B, continuing SoC-CT without SBRT.

Arm A: The primary tumor is treated with SBRT (6.6 Gy x 5) on a MR-LINAC in breath-hold technique. This scheme was shown to have a reasonable toxicity profile on a conventional LINAC. A low toxicity profile is even more important in patients with metastatic and therefore definitively incurable cancer. Therefore, treatment is performed on a MR-LINAC to deliver high doses to the tumor while keeping the toxicity profile as low as possible. For this purpose, daily adaptive planning is performed aiming to maintain stringent dose constraints for organs at risk (duodenum / stomach / bowel / kidney). Chemotherapy will be continued after SBRT. Arm B: Continuing SoC-CT (according to clinical routine appr. 2 weeks after the previous cycle) without SBRT.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with histologically proven, metastatic pancreatic adenocarcinoma of the pancreatic head or body amenable for MR-guided adaptive SBRT with at least stable disease after 8 weeks of standard of care doublet chemotherapy
* age >18 years
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0, 1 or 2
* Ability to follow study instructions and likely to attend and complete all required visits

Exclusion Criteria:

* Subjects not able to give consent
* Subjects without legal capacity who are unable to understand the nature, scope, significance and consequences of this clinical study
* Simultaneous participation in another clinical study or participation in any clinical trial involving an investigational medicinal product or treatment within 30 days prior to beginning of this study
* Subjects with a physical or psychiatric condition which at the investigator's discretion may put the subject at risk, may confound the study results, or may interfere with the subject's participation in this study
* Women of child bearing potential or sexually active males not willing to use effective contraception while on treatment and 12 weeks after the end of treatment (such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices) unless they are surgically sterilized / hysterectomized or there are any other criteria considered sufficiently reliable by the investigator in individual cases
* Biopsy proven tumor invasion into the stomach and/or duodenum
* Medically uncontrolled pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2025-11-11 (Actual); Study Completion 2025-11-11 (Actual)

PRIMARY OUTCOMES:
Mean cumulative pain index | through study completion, at least 24 weeks or until death
  Mean Cumulative pain index: AUC of pain scores rated every 4 weeks until death or end of study using numeric rating scale (NRS, 0= no pain, 10 = worst pain) divided by number of multiples of 4 weeks since randomization

SECONDARY OUTCOMES:
Number of biliary complications | through study completion, at least 24 weeks or until death
  Biliary complications defined as cholangitis or post-hepatic cholestasis requiring drainage
Malnutrition | through study completion, at least 24 weeks or until death
  Nutritional status measuring bioimpedance-derived phase angle (BIA) every 12 weeks
Treatment toxicity | through study completion, at least 24 weeks or until death
  Treatment toxicity according to CTCAE v5.0
Death from any cause | through study completion

CONTACTS AND LOCATIONS:
Overall Officials: Maximilian Niyazi, Prof. Dr., Principal Investigator — Depatment of Radiation Oncology, University Hospital, LMU Munich
Locations (3):
- Germany (2):
  - University of Munich, Dep. of Radiation Oncology, Munich, Bavaria
  - University Hospital of Heidelberg, Dep. of Radiation Oncology, Heidelberg
- University Hospital of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pavic M, Niyazi M, Wilke L, Corradini S, Vornhulz M, Mansmann U, Al Tawil A, Fritsch R, Horner-Rieber J, Debus J, Guckenberger M, Belka C, Mayerle J, Beyer G. MR-guided adaptive stereotactic body radiotherapy (SBRT) of primary tumor for pain control in metastatic pancreatic ductal adenocarcinoma (mPDAC): an open randomized, multicentric, parallel group clinical trial (MASPAC). Radiat Oncol. 2022 Jan 25;17(1):18. doi: 10.1186/s13014-022-01988-6. PMID 35078490